CLINICAL TRIAL: NCT05697224
Title: Role of Aschistosoma Haematobiumspecific microRNAas Atumor Marker for Early Diagnosis and Prognosis of Bilharzial Bladder Cancer in Eygpt
Brief Title: Aschistosoma Haematobiumspecific microRNAas a Tumor Marker for Early Diagnosis and Prognosis of Bilharzial Bladder Cancer in Eygpt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Omar Ali, assistant lecturar at parasitology department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-med-22-11-12
Record Dates: First submitted 2023-01-15; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronicurinary schistosomiasis (Active Comparator)
  Interventions: Diagnostic Test: urinary micro RNA detection
- bladder cancer diseased patients (Active Comparator)
  Interventions: Diagnostic Test: urinary micro RNA detection

INTERVENTIONS:
Diagnostic Test: urinary micro RNA detection — Urinary Sha-miR-71a gene expression analysis Total RNA extraction and purification Sha-miR_71a gene expression analysis MAPK-3 gene expression analysis

SUMMARY:
miRNAs have been detected in different bodily fluids, which suggests significant potential, such as their use as biomarkers in diagnostics and prognostics. Sha-mir-71a was abundantly found in the urine of patients with bladder cancer as compared to benign bladder cystitis associated with schistosomiasis . Additionally, this miRNA was more highly detected in urine samples from patients with bilharzial bladder cancer than bladder cancer not associated with bilharziasis (schistosomiasis), suggesting its specificity in the identification of bladder cancer associated with infection.

ELIGIBILITY:
Inclusion Criteria:

* urinary symptoms (hematuria, urinary retention, dysuria… etc.), who were planned to undergo cystoscopy for suspicion of bladder cancer (BC) or benign bilharzial cystitis (Bil), will be selected.

Exclusion Criteria:

* : In bladder cancer group Patients who have received chemotherapy, or with previously diagnosed other malignancy within the past 5 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
use micro RNAas adiagnostic test for early diagnosis of shistosomal bladder cancer | one year
  Sha-mir-71a could be a biomarker with diagnostic and prognostic value

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Eissa S, Matboli M, Essawy NO, Kotb YM. Integrative functional genetic-epigenetic approach for selecting genes as urine biomarkers for bladder cancer diagnosis. Tumour Biol. 2015 Dec;36(12):9545-52. doi: 10.1007/s13277-015-3722-6. Epub 2015 Jul 3. PMID 26138586
- [Background] Abd El-Aal AA, Bayoumy IR, Basyoni MM, Abd El-Aal AA, Emran AM, Abd El-Tawab MS, Badawi MA, Zalat RM, Diab TM. Genomic instability in complicated and uncomplicated Egyptian schistosomiasis haematobium patients. Mol Cytogenet. 2015 Jan 22;8(1):1. doi: 10.1186/s13039-014-0104-5. eCollection 2015. PMID 25628757
- [Background] Chen L, Yuan L, Wang G, Cao R, Peng J, Shu B, Qian G, Wang X, Xiao Y. Identification and bioinformatics analysis of miRNAs associated with human muscle invasive bladder cancer. Mol Med Rep. 2017 Dec;16(6):8709-8720. doi: 10.3892/mmr.2017.7726. Epub 2017 Oct 4. PMID 28990088